CLINICAL TRIAL: NCT01089894
Title: Clinical Application of 18F-FLT PET in Lung Tumors
Brief Title: Clinical Application of 18F-3'-Fluoro-3'-Deoxy-L-thymidine (18F-FLT) Positron Emission Tomography (PET) in Lung Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yen RF, National Taiwan University Hospital
Other Study IDs: 200712071R
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer
Keywords: 18F-FLT; PET; non-small cell lung cancer; cell proliferation; therapeutic response; 18F-3'-fluoro-3'-deoxy-L-thymidine (18F-FLT)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 18F-FLT 1: 18F-FLT in differentiating benign from malignant pulmonary nodules
- 18F-FLT 2: 18F-FLT in evaluating therapeutic response of platinum-based chemotherapy (The chemotherapeutic drugs used in the study are all approved by the Department of Health, Taiwan.)
- 18F-FLT 3: 18F-FLT in evaluating therapeutic response of EGFR tyrosin kinase inhibitors (The target therapeutic drugs used in the study are all approved by the Department of Health, Taiwan.)

SUMMARY:
The ability of 18F-FDG PET for characterizing lung nodule remains a challenge, especially in Taiwan where tuberculosis is still prevalent.

18F-3'-fluoro-3'-deoxy-L-thymidine (18F-FLT), a radiolabeled analog of thymidine, can be trapped within the cytosol after being monophosphorylated by thymidine kinase-1 (TK-1), a principle enzyme in the salvage pathway of DNA synthesis. It has been demonstrated in cell culture, animal models and clinical studies that the accumulation of 18F-FLT is closely associated with cellular proliferation. 18F-FLT PET may be more accurate than 18F-FDG PET in differentiating benign from malignant pulmonary lesions. In addition, the correlation between 18F-FLT uptake and cellular proliferation hints the usefulness of 18F-FLT PET for monitoring treatment response with cytostatic anticancer drugs.

We thus design this prospective 3-year project

1. To evaluate the usefulness of 18F-FLT PET and 18F-FDG PET in differentiating benign from malignant pulmonary nodules in Taiwan where tuberculosis is still prevalent.
2. To assess the usefulness of 18F-FLT PET in early prediction of therapeutic response of platinum-based chemotherapies or EGFR inhibitors for NSCLC patients.
3. To correlate 18F-FLT uptake with EGFR mutation status, therapeutic response and survival for NSCLC patients.

DETAILED DESCRIPTION:
Lung cancer has become a leading cause of cancer death in Taiwan. 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET) using has been found to be effective in diagnosing, staging, and restaging primary non-small cell lung cancer (NSCLC). However, 18F-FDG is not tumor specific. It may also show increased uptake in benign tumors and tissue with inflammatory cells, such as macrophages and fibroblast. Therefore, the ability of 18F-FDG PET for characterizing lung nodule remains a challenge, especially in Taiwan where tuberculosis is still prevalent.

Recently, 18F-3'-fluoro-3'-deoxy-L-thymidine (18F-FLT), a radiolabeled analog of thymidine, has been synthesized for imaging tumor cell proliferation in vivo. The tracer is trapped within the cytosol after being monophosphorylated by thymidine kinase-1 (TK-1), a principle enzyme in the salvage pathway of DNA synthesis. It has been demonstrated in cell culture, animal models and clinical studies that the accumulation of 18F-FLT is dependent on the presence of TK-1 and therefore is closely associated with cellular proliferation. Malignant lung lesions revealed significant 18F-FLT accumulation while benign lung tumors showed no 18F-FLT uptake. Therefore, 18F-FLT PET may be more accurate than 18F-FDG PET in differentiating benign from malignant pulmonary lesions. In addition, the correlation between 18F-FLT uptake and cellular proliferation hints the usefulness of 18F-FLT PET for monitoring treatment response with cytostatic anticancer drugs.

In the meantime, the cyclotron and hot lab facility in National Taiwan University Hospital (NTUH) has developed 18F-FLT successfully. After careful quality assurance and animal experiments, it is now ready to perform clinical studies on human beings.

We thus design this prospective 3-year project

1. To evaluate the usefulness of 18F-FLT PET and 18F-FDG PET in differentiating benign from malignant pulmonary nodules in Taiwan where tuberculosis is still prevalent.
2. To assess the usefulness of 18F-FLT PET in early prediction of therapeutic response of platinum-based chemotherapies or EGFR inhibitors for NSCLC patients.
3. To correlate 18F-FLT uptake with EGFR mutation status, therapeutic response and survival for NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

18F-FLT 1:

1. indeterminate pulmonary nodule(s)
2. has been scheduled an 18F-FDG PET for characterization of their indeterminate pulmonary nodule(s)
3. consent to perform an additional 18F-FLT PET
4. will receive biopsy or surgery for the pulmonary nodule(s)

18F-FLT 2:

1. has pathological proved NSCLC
2. is staged as inoperable advanced NSCLC
3. has been scheduled to receive platinum-based chemotherapy
4. consents to received 18F-FLT PET studies before, at the day before initiation of 2nd cycle of therapy or at 7 days after completion of therapy

18F-FLT 3:

1. has pathological proved NSCLC
2. is staged as inoperable advanced NSCLC
3. has been scheduled to receive EGFR tyrosine kinase inhibitor therapy
4. consents to received 18F-FLT PET studies before, at the 2nd day or at the 7th day of therapy
5. consents to undergo EGFR mutation analysis

Exclusion Criteria:

1. Patients with other known malignancies
2. Age under 18 years
3. Hematological parameters: WBC < 3000/L or platelet < 75,000/L (WHO toxicity criteria of grade 1)
4. Abnormal liver function: AST or ALT > 78U/L (WHO toxicity criteria of grade 1)
5. Renal function: Creatinine > 2.0 mg/dl (WHO toxicity criteria of grade 1)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18F-FLT 1: 18F-FLT in differentiating benign from malignant pulmonary nodules
  18F-FLT 2: 18F-FLT in evaluating therapeutic response of platinum-based chemotherapy (The chemotherapeutic drugs used in the study are all approved by the Department of Health
  18F-FLT 3: 18F-FLT in evaluating therapeutic response of EGFR tyrosin kinase inhibitors (The target therapeutic drugs used in the study are all approved by the Department of Health, Taiwan.)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruoh-Fang Yen, M.D PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan